CLINICAL TRIAL: NCT00081549
Title: A Phase I/II Study of Aroplatin and Gemcitabine In Subjects With Unresectable, Locally Advanced And/Or Metastatic Pancreatic Cancer
Brief Title: Aroplatin and Gemcitabine in Patients With Advanced Pancreatic Cancer Resistant to Standard Therapies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aronex Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C-726-02
Record Dates: First submitted 2004-04-15; First posted 2004-04-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Cancer; Neoplasms Pancreatic; Pancreas Cancer; Pancreas Neoplasms; Pancreatic Tumor; Pancreas Tumor; Unresectable; Metastatic; Refractory
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — bis-neodecanoato-1,2-diaminocyclohexaneplatinum(II)

INTERVENTIONS:
Drug: Aroplatin (Liposomal NDDP, L-NDDP)

SUMMARY:
This study is a Phase I/II study. In Phase I of this study, the objective is to determine the maximum tolerated dose (MTD) of combination therapy with Aroplatin and gemcitabine (Gemzar®) in subjects with unresectable, locally advanced and/or metastatic pancreatic cancer. In Phase II, the primary objective is to evaluate survival after therapy with Aroplatin and gemcitabine at the identified MTD in subjects with unresectable, locally advanced and/or metastatic pancreatic cancer. Secondary objectives are to evaluate the severity and quantity of adverse events and determine the proportion of non-progressors and the progression-free interval.

DETAILED DESCRIPTION:
Phase I Primary Objective:

* Determine the maximum tolerated dose (MTD) of combination therapy with Aroplatin and gemcitabine (Gemzar®) in subjects with unresectable, locally advanced and/or metastatic pancreatic cancer.

Phase II Primary Objective:

* Evaluate survival after therapy with Aroplatin and gemcitabine at the MTD in subjects with unresectable, locally advanced and/or metastatic pancreatic cancer.

Phase II Secondary Objective:

* Evaluate the severity and quantity of adverse events and determine the proportion of non-progressors and the progression-free interval.

ELIGIBILITY:
Inclusion Criteria

* Pancreatic cancer (AJCC Stage II-IV);
* Unresectable cancer;
* Measurable disease (RECIST criteria);
* No prior therapy;
* ECOG Score 0-2
* Life expectancy greater then or equal to three months;
* Adequate hematopoietic, liver and renal function;
* Women of child-bearing potential must have negative urine/serum pregnancy test;
* Signed written informed consent;
* Subjects must be willing to be followed during the course of the treatment/observation and follow-up.

Exclusion Criteria:

* Prior therapy for pancreatic cancer;
* Previously diagnosed brain metastases if symptomatic and requiring active therapy;
* Other cancers within the last five years, with the exception of adequately treated cone-biopsied in-situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin;
* Any serious concomitant medical or mental illness requiring intense therapy and interfering with participation in this study
* Primary or secondary immunodeficiency, or use of corticosteroids immunosuppressive medication;
* Women must not be pregnant or breast-feeding;
* Participation in any clinical trial involving investigational drugs within one month from enrollment into the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111